CLINICAL TRIAL: NCT04437927
Title: Impact of 100mL Lipid Emulsion for Intravenous for Suppression of Myocardial Glucose
Brief Title: Impact of 100mL Lipid Emulsion for Intravenous for Suppression of Myocardial Glucose Metabolism in 18F-FDG PET/CT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: 20-11
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-06

CONDITIONS: Metabolic Preparation; Myocardial Inflammation
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective patients: 30 consecutive patients with cardiac FDG PET prescribed
- Control: 30 patients referred for cardiac FDG PET in the nuclear medicine department of the Centre Hospitalier Princesse Grace

SUMMARY:
There is increasing evidence that [18F]-2-fluoro-2-deoxy-D-glucose (18F-FDG) PET/CT is useful in the identification and treatment of disease processes that involve cardiac inflammation and infection. Current applications include imaging intra-cardiac device and prosthetic valve infections, evaluating patients with known or suspected cardiac sarcoidosis or other inflammatory cardiomyopathies.

However, because normal myocardium can metabolize both glucose and free fatty acids (FFAs), physiological accumulation of FDG in the myocardium can interfere with the recognition of abnormal FDG uptake.

The use of a low-carbohydrate diet with a prolonged fast ≥ 12 h nutrition followed by a fast of at least four hours is the effective preparation recommended to suppress physiological myocardial FDG uptake.

However, the rate of suppression of physiological accumulation of FDG with this method in our center is only 50%.

DETAILED DESCRIPTION:
Methodology :

Group of 30 consecutive patients with cardiac FDG PET prescribed, prospectively enrolled, compared to a group with the last 30 patients referred for cardiac FDG PET in the nuclear medicine department of the Centre Hospitalier Princesse Grace.

Procedures :

Infusion of 100mL lipid emulsion for intravenous two hours before cardiac FDG PET/CT:

* Infusion rate will be 20 mL/hour during the initial 10 minutes (3 mL Intralipid)
* The dose will be then increased to 40 mL/hour for the next 10 minutes (6 mL Intralipid)
* Finally, for the next 50 minutes the dose will be increased to 100 mL/hour (83mL Intralipid)

ELIGIBILITY:
Inclusion Criteria:

* Patients with an FDG PET/CT prescribed to explore cardiac disease process

Exclusion Criteria:

* renal insufficiency,
* uncompensated diabetes mellitus,
* pancreatitis,
* liver insufficiency,
* hypothyroidism
* metabolic disorders
* sepsis.
* soy protein allergy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group of 30 consecutive patients with cardiac FDG PET prescribed, prospectively enrolled, compared to a group with the last 30 patients referred for cardiac FDG PET.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Uptake in the heart scoring according to a visual scale | day 1
  * Score of 0: complete myocardial suppression
  * Score of 1: incomplete myocardial suppression with increased myocardial FDG uptake hampering myocardial interpretation but not cardiac valves.
  * Score of 2: incomplete myocardial suppression with increased myocardial FDG uptake hampering myocardial and mitral or aortic valve interpretations.
  * Score of 3: incomplete myocardial suppression with increased myocardial FDG uptake hampering myocardial and both mitral and aortic valves interpretations.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

REFERENCES:
- [Derived] Dietz M, Paulmier B, Berthier F, Civaia F, Mocquot F, Serrano B, Nataf V, Hugonnet F, Faraggi M. An Intravenous 100-mL Lipid Emulsion Infusion Dramatically Improves Myocardial Glucose Metabolism Extinction in Cardiac FDG PET Clinical Practice. Clin Nucl Med. 2021 Jun 1;46(6):e317-e324. doi: 10.1097/RLU.0000000000003556. PMID 33630808